CLINICAL TRIAL: NCT02086058
Title: Gene Expression in the Bladder in Children With an Overactive Bladder and Daytime Urinary Incontinence
Brief Title: Gene Expression in the Overactive Bladder in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: GeneOAB
Record Dates: First submitted 2014-03-06; First posted 2014-03-13 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Overactive Bladder; Children
Keywords: overactive bladder; daytime urinary incontinence; children; gene expression
MeSH Terms: conditions — Urinary Bladder, Overactive; Diurnal Enuresis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bladder biopsies from the back-wall og the bladder.
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study (the hypothesis) is to identify differences in the gene expression profile in the bladder muscle and hereby gain greater knowledge about the muscular mechanisms that cause overactive bladder and daytime urinary incontinence in children older than 5 years. A secondary aim is to examine how this gene expression profile differs from children with a neurogenic overactive bladder and how the gene expression profile changes from childhood till adulthood. Such new knowledge will result in a more precisely targeted and hence effective treatment of overactive bladder.

The results will be obtained by retrieving bladder biopsies from children and adults suffering from an overactive bladder or a neurogenic bladder. These biopsies will undergo molecular analysis and the investigators will compare them with biopises from bladder healthy adults and children.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Group 1 (non-neurogenic bladder/overactive bladder):

* age 5-14 years of age
* patients must have filled out 48-hour bladder diaries
* a minimum of 4 micturitions per day (assessed from the bladder diaries)
* functional daytime urinary incontinence
* overactive bladder as defined by urgency
* no signs of neurogenic bladder dysfunction on invasive urodynamics
* a non-remarkable clinical examination
* normal BMI (between 3-97 percentile)
* informed oral and written consent from the child and both parents/legal guardian. In the informed consent the parents /legal guardian have given permission to the authorities (The Danish Ethical Committee), so that they may get information about the child during monitoring and quality inspection visits.
* no effect of prior treatment of at least 6 months urotherapy
* no effect of prior treatment of at least 3 months of anticholinergic treatment
* planned to undergo a cystoscopy under anesthesia

Group 2:

* 5-14 years of age or >18 years old
* diagnosed with a neurogenic bladder (i.e. caused by myelomeningocele)
* informed oral and written consent from the child and both parents/legal guardian. In the informed consent the parents /legal guardian have given permission to the authorities (The Danish Ethical Committee), so that they may get information about the child during monitoring and quality inspection visits.
* planned to undergo a cystoscopy under anesthesia

Group 3:

* age 5-14 years of age or >18 years old
* a non-remarkable clinical examination
* a normal voiding pattern
* a minimum of 3 micturitions per day
* planned to undergo a cystoscopy under anesthesia

Exclusion Criteria:

Group 1:

* Neurological and/or anatomical abnormalities in the lower urinary tract
* a medical history, clinical or biochemical tests that indicate that the child suffers from any type of disease (such as acute urinary infection or diabetes) or condition (such as pregnancy) influencing the child´s possibility of participating in the study, or that may effect the study parameters that are under examination.
* ongoing fecal problems such as fecal incontinence or constipation
* prior surgery involving the bladder
* ongoing urinary tract infections
* ongoing treatment with any type of medicine that may effect the study parameters that are under examination

Group 2:

* a medical history, clinical or biochemical tests that indicate that the child suffers from any type of diseases (such as diabetes) or conditions (such as pregnancy) influencing the child´s possibility of participating in the study, or that may affect the study parameters that are under examination.
* ongoing treatment with any type of medicine that may affect the study parameters that are under examination

Group 3:

* Neurological and/or anatomical abnormalities in the lower urinary tract
* urinary incontinence and an overactive bladder with urinary incontinence
* a medical history, clinical or biochemical tests that indicate that the patient suffers from any type of disease (such as acute urinary tract infection or diabetes) or condition (such as pregnancy) influencing the patient´s possibility of participating in the study, or that may effect the study parameters that are under examination.
* any type of bladder disease or any disease secondary affecting the bladder
* prior bladder surgery
* ongoing urinary tract infection
* ongoing treatment with any type of medicine that may effect the study parameters that are under examination.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will include 3 groups of patients Group 1: children with an overactive bladder and daytime urinary incontinence Group 2: Children and adults with a neurogenic bladder Group 3: children and adults who have a healthy bladder
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-09 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Up- and down regulation of genes expressed in the bladder | collection of bladder material and analysis will take approximately 2 years
  We will evaluate the gene expression (which genes are up- and/or down regulated) in the bladder in healthy children compared to children suffering from an overactive bladder. This gene expression will then be compared to the gene expression in bladder tissue from adults, to evaluate what happens in the bladder from childhood to adulthood.

CONTACTS AND LOCATIONS:
Overall Officials: Luise Borch, M.D, Principal Investigator — University of Aarhus
Locations (1):
- Center for child incontinence, Aarhus University hospital, Aarhus, Aarhus N, Denmark